CLINICAL TRIAL: NCT04457388
Title: Tele- Yoga Therapy for Patients With Chronic Pain During Covid-19 Lockdown: A Prospective Non-randomized Single Arm Clinical Trial
Brief Title: Tele-Yoga Therapy for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarogyam UK (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AU/018
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Chronic Pain
Keywords: Tele-Yoga Therapy; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tele-Yoga Therapy (Experimental): Individualised Yoga therapy based on participant's clinical condition and personal needs. Twice a week sessions were carried out by trained and experienced Yoga therapist via video conference with each therapy for individualized based on each participant.
  Interventions: Other: Tele-Yoga Therapy

INTERVENTIONS:
Other: Tele-Yoga Therapy — Yoga practices combining with joint loosening exercises (Sukshma Vyayama), postures (Asana), breathing exercises (Pranayama), relaxation techniques and chanting ( A, U, M, and AUM { ૐ}) syllable chants meditation. Each session ended with home practice exercises given to the participants to practice everyday.

SUMMARY:
Chronic pain is highly prevalent and associated with a large symptom burden, that is had been more concerning during Covid-19 outbreak and lockdown. Benefits of yoga in chronic pain management are very well known. With this background we developed Tele-Yoga therapy program and evaluated the success of this single arm study.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain for at least 3 months
* Having access to internet and video calls

Exclusion Criteria:

* Pregnant or breast-feeding women,
* Patients not willing to give written consent
* Patients with severe psychiatric or personality disorder
* Malignancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | From baseline to 6-week post intervention
  visual-analogic scale (VAS), using pain level from "no pain" (0) to "worst imaginable pain" (10)

SECONDARY OUTCOMES:
Pain Disability | From baseline to 6-week post intervention
  Pain Disability Index (PDI) using seven rating scales, structured in Likert form, from "no disability" (0) to "worst disability" (10)
Anxiety | From Baseline to 6-week post intervention
  Hospital Anxiety Depression Scale, consisting of 7 scales for measuring anxiety levels
Depression | From baseline to 6-week post intervention
  Hospital Anxiety Depression Scale, consisting of 7 scales for measuring depression levels

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, Principal Investigator — Aarogyam UK; Dipa Modi, Study Chair — Aarogyam UK; Bhavna Pandya, Study Chair — Aarogyam UK
Locations (1):
- Aarogyam UK, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided